CLINICAL TRIAL: NCT05286502
Title: NW500 Non-Mydriatic Retinal Camera Clinical Performance Study
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THS-TPCN-2022-001
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-03

CONDITIONS: Fundus Photography
MeSH Terms: interventions — Fluorescein Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults 18 years old or older
  Interventions: Device: fundus photography

INTERVENTIONS:
Device: fundus photography — color fundus photography

SUMMARY:
Comparison of color fundus images acquired by the Topcon NW500 non-mydriatic retinal camera (investigational device) and the Topcon TRC-NW400 (predicate device)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age or older on the date of informed consent.
* Subjects who are able to understand the written informed consent and are willing to participate as evidenced by signing the informed consent.

Exclusion Criteria:

* Subjects who are unable to tolerate ophthalmic imaging.
* Subjects with poor fixation or ocular media not sufficiently clear to obtain acceptable images.
* Subjects who cannot follow instructions to complete the required testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years old or older.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
fundus photo image quality | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Topcon Healthcare Solutions, Oakland, New Jersey, United States